CLINICAL TRIAL: NCT03705403
Title: Stereotactic Ablative Body Radiotherapy (SABR) Combined with Immunotherapy (L19-IL2) in Stage IV NSCLC Patients, ImmunoSABR: a Multicentre, Randomised Controlled Open-label Phase II Trial
Brief Title: IMMUNOtherapy and Stereotactic ABlative Radiotherapy (IMMUNOSABR) a Phase II Study
Acronym: IMMUNOSABR2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial is not transitioning to the Clinical Trial Regulation (CTR) EU No 536/2014.
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other); The Netherlands Cancer Institute (Other); University Medical Center Nijmegen (Other); Erasmus Medical Center (Other); University Ghent (Other); KU Leuven (Other); Centre Oscar Lambret (Other); Gasthuis Zusters Antwerpen (Other); University College, London (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University Hospital Dresden (Other); University Hospital Tuebingen (Other); Heidelberg University (Other); Catholic University of the Sacred Heart (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UM2018IMMUNOSABR2RLPL
Record Dates: First submitted 2018-06-27; First posted 2018-10-15 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: NSCLC Stage IV; Metastatic Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — L19-IL2 immunocytokine; Radiation; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This will be a multicentre, randomised controlled open-label phase II trial testing if the combination of (SAB)R and immunocytokine L19-IL2 improves the progression-free survival in patients with limited metastatic non-small cell lung cancer (NSCLC). The patients included in the trial will be stratified for the metastatic load (oligo; max 5 or diffuse; 6-10 metastases). After randomisation, patients will be assigned either to the experimental arm or the standard of care (SOC) arm. Depending on the metastatic load, patients with (max 5 metastases) will receive in the experimental arm SABR to all lesions followed by L19-IL2 followed by standard of care therapy. Patients with more extensive metastatic disease (6 to up to 10 metastasis) in the experimental arm will be included following first or second line treatment with a platinum doublet and receive radiotherapy (3x8 Gy) to at least one (symptomatic) lesion, followed by L19-IL2 followed by SOC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Standard of Care (SOC) according to the local and national guidelines: (wait and see or surgery and/or chemotherapy and/or standard (symptomatic) radiation therapy and/or SABR (oligometastatic disease)
  Interventions: Radiation: Radiation
- Experimental treatment (Experimental): Standard of Care (SOC SABR (oligometastatic disease) or radiation therapy (diffuse disease) + L19-IL2 up to 6 cycles (Darleukin)
  Interventions: Drug: Darleukin; Radiation: Radiation

INTERVENTIONS:
Drug: Darleukin — The product name refers to the molecule structure, in fact, L19-IL2 is a recombinant fusion protein composed of two moieties: L19, a human monoclonal antibody fragment in the single chain Fv (scFv) format, bound via a flexible linker to IL2, the human cytokine Interleukin-2.
  Other Names: L19 - IL2
  Arms: Experimental treatment
Radiation: Radiation — Radiotherapy
  Other Names: Radiotherapy

SUMMARY:
This will be a phase II trial testing if the combination of stereotactic ablative body radiotherapy (SABR) and L19-IL2 improve the progression-free survival in patients with limited metastatic non-small cell lung cancer (NSCLC). The trial consists of one cohort with two arms; C-arm and an E-arm.

Patients with oligometastatic disease will receive SABR to minimal 1 and max all metastatic sites (max 5 sites irradiated) and patients with diffuse metastatic lesions (6 to max 10) will receive radiotherapy to max 5 sites. In the experimental arm, immunotherapy will be given after irradiation.

DETAILED DESCRIPTION:
IMMUNOSABR will include 126 patients. In this single-stage controlled randomised open-label phase II trial, we aim to demonstrate an absolute increase in progression-free survival (primary endpoint). PFS will be determined as the time between randomisation and disease progression, according to RECIST 1.1, death due to any cause or last patient contact alive and progression-free. Patients will be randomized between control (no immunocytokine) and experimental arms (with immunocytokine L19-IL2) in a 1:1 ratio. The accrual period will be 29 months (or 2.41 years), and the minimum follow-up will be 18 months (or 1.5 years), making the total study duration 47 months. Comparison between control and experimental arms will be made using the Log-Rank statistic. This test for superiority will be one-sided with the desired type I error of 0.10 and power of 0.90.

Patients enrolled in the trial will be randomised into the control arm (C-arm) or experimental arm (E-arm).

* C-arm: Standard of Care (SOC) according to the local and national guidelines: (wait and see or surgery and/or chemotherapy and/or standard (symptomatic) radiotherapy and/or SABR, oligometastatic disease.
* E-arm: SABR (oligometastatic disease) or radiotherapy (diffuse disease) + L19-IL2 up to 6 cycles (+ aPD(L)1 if SOC)

The expected 1.5-year PFS is 15% in the C-arm and 35% in the E-arm. A sample size of 116 patients (58 patients per treatment arm) is needed to show this difference of 20% in PFS, using a logrank test with a two-sided alpha of 0.05 and power of 85%. Patients will be evenly divided over the two arms. Assuming a drop-out rate of 10%, a total of 126 patients (63 per arm) need to be included.

Primary objective The main objective of the trial is to test if the activity of the combination of (SAB)R and L19-IL2 in patients with metastatic NSCLC will result in improved progression-free survival (PFS) compared to the SOC.

Secondary Objectives

* Assessment of the PFS of the patient cohort, at 5 years after randomisation.
* Assessment of the overall survival of the patient cohort, at 5 years after randomisation.
* To assess the toxicity of this treatment schedule;
* To assess Quality of Life (QoL);
* To assess the occurrence of an Out of Field Radio-Immune (OFRI) response / abscopal effect using imaging;
* To assess the occurrence of an In Field Radio-Immune (IFRI) response using imaging;
* To perform correlative biomarker studies related to treatment response.

Exploratory endpoints:

* Correlative biomarker studies:

  * Tumour tissue: e.g EDB expression, non-synonymous mutations, immune monitoring;
  * Blood: e.g. EDB expression, cfDNA, and immune monitoring;
  * Radiomics on CT and if available MRI;
  * Faeces: diversity in microbiota.
* iRECIST
* Tumour grow kinetics

ELIGIBILITY:
Inclusion criteria

Oligometastatic disease (≤5 metastases)

* Histological confirmed limited metastatic adult NSCLC patients, regardless of the PD-L1 status.

  * Maximum of 5 metastatic lesions, maximum two brain lesion with a total cumulative diameter of 5cm is allowed.

SOC baseline imaging e.g MRI and/or PET-CT and CT-brain or MRI brain and/or CT-scan with at least covering thorax-upper abdomen-brain, within 6 weeks prior to randomisation.

If a patient has unclear lesions in the liver or brain an MRI would be advised following the ESMO guidelines.

o In patients with 2 lung tumours, it can be unclear if the patient has 2 concurrent primary tumours or a primary lung tumour with 1 metastasis. In this case, the local multidisciplinary tumour board will decide whether the patient has an M1 disease or not.

• Previous treatment: Prior cancer treatments are allowed but must be discontinued for at least 4 weeks before randomisation. In case of maintenance chemotherapy, this therapy will only be started after the end of the L19-IL2 treatment or only in case of Anti-PD(L)1 treatment, during L19-IL2 therapy.

* Age of 18 years or older.
* WHO performance status 0-1;
* Adequate bone marrow function, evaluated in the local laboratory (Lab): Absolute Neutrophil Count (ANC) of ≥ 1.0 x 109 /L, platelet count ≥ 100 x 109/L, Haemoglobin (Hb) ≥ 6.0 mmol/L (or 9.67 g/dL) (it is allowed to give a blood transfusion if Hb is initially too low);
* Adequate hepatic function (evaluated in the local lab): total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution or ≤ 5 in case of liver metastasis);
* Adequate renal function (evaluated in the local lab): creatinine clearance of at least 40 ml/min;
* Adequate endocrine (TSH, FT4) function, local guidelines
* The patient is capable of complying with study procedures;
* Life expectancy of at least 12 weeks;
* Negative serum pregnancy test for females of childbearing potential.
* Signed and dated written informed consent.
* Ability to comply with contraception requirements:

Non-sterilised, sexually active male patient with a female partner who is of child-bearing age, must use two acceptable birth control methods like a condom combined with spermicidal cream or gel from the first dose of study medicine, during the study and at least up to 12 weeks after the last administration of the study medicine and up to 5 months after the last dose of the medicine with anti-PDL)1 as an action mechanism (if you get this product besides the study medicine), as an addition to the use, by the female partner, of as described in the following section:

Women of childbearing potential (WOCBP) and WOCBP partners of male patients must be using, from the screening to three months following the last study drug administration and 4 5 months after last dose of anti-PD(L)1 maintenance treatment, effective contraception methods ((a) IUD (IUD) or intrauterine hormone delivery system (IUS), b) combined (with estrogen and progesterone) hormonal contraception associated with ovulation inhibition (oral, intravaginal, transdermal), c) hormonal contraception with progesterone only associated with ovulation inhibition (oral, injectable, implantable), as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html).

Poly-metastatic disease (6 to 10 metastases)

• Histological confirmed limited metastatic adult NSCLC patients, regardless of the PD-L1 status.

A minimum of 6 and maximum of 10 metastatic lesions, maximum two brain lesion with a total cumulative diameter of 5cm is allowed.

At least one measurable lesion (according to RECIST 1.1) that has no overlap with the PTV of the lesion subjected to radiotherapy.

• Previous treatment: The time between the last administration of chemotherapy and the randomisation must be at least 4 weeks. In case of maintenance chemotherapy, this therapy will only be started after the study if e-arm, allowed during c-arm. In case of Anti-PD(L)1 treatment, this is allowed in both arms, so also during L19-IL2 therapy.

* Age of 18 years or older;
* WHO performance status 0-1;
* Adequate bone marrow function (evaluated in the local lab): Absolute Neutrophil Count (ANC) of ≥ 1.0 x 109 /L, platelet count ≥ 100 x 109/L, Hb ≥ 6.0 mmol/L (or 9.67 g/dL) (it is allowed to give a blood transfusion if Hb is initially too low);
* Adequate hepatic function (evaluated in the local lab): total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution or ≤ 5 in case of liver metastasis);
* Adequate renal function (evaluated in the local lab): creatinine clearance of at least 40 ml/min;
* Adequate endocrine (TSH, FT4) function, local guidelines;
* The patient is capable of complying with study procedures;
* Life expectancy of at least 12 weeks;
* Negative serum pregnancy test for females of childbearing potential;
* Ability to comply with contraception requirements (see oligo)
* Signed and dated written informed consent.

Exclusion criteria

* More than 10 metastatic lesions.
* More than 2 brain metastatic lesions.
* 2 brain metastases with a cumulative diameter larger than 5 cm.
* Patients with non-infectious pneumonitis, uncontrolled thyroid disease, pleuritis, pericarditis and peritonitis carcinomatosis.
* Patients who received live vaccines 30 days or fewer prior to enrolment.
* Patients who are already actively participating in another study.
* Patients who need simultaneous radiation on the primary tumour and metastatic lesion(s). For these patients it might be an option to treat the primary tumour first although this is not mandatory for this study. There must be minimal four weeks between last treatment and randomisation.
* Whole brain radiotherapy (WBRT) is not allowed, although it is accepted when given at least 4 weeks prior to randomisation or after the treatment period. Patients with stable brain metastases are not excluded.
* Previous radiotherapy to an area that would be re-treated by (SAB)R, resulting in overlap of the high dose areas.
* Maintenance therapy with Anti-PD(L)1 treatment combined with chemotherapy is not allowed during treatment ((SAB)R and L19-IL2 cycles).
* Other active malignancy or malignancy within the last 2 years (except localised skin basal/squamous cell carcinoma, non-muscle invasive carcinoma of the bladder or in situ carcinoma from any site).
* Concomitantly administered glucocorticoids may decrease the activity of IL2 and therefore should be avoided. However, patients who develop life-threatening signs or symptoms may be treated with dexamethasone until toxicity resolves or reduces to an acceptable level (generally grade 1 and 2, however must be based at the research physician's discretion).
* History of allergy to intravenously administered proteins/peptides/antibodies/ radiographic contrast media.
* HIV positive; active HIV infection, or active hepatitis B or C (assessed in local lab).
* Systemic treatment with either corticosteroid (>10 mg daily prednisone equivalents) or Interferon alpha or immunosuppressive medications within 14 days prior to randomisation. Topical or inhalation steroids are allowed. If a patient needs to take unexpectedly immunosuppressive medication during the trial, it will be allowed but decreasing the dose as soon as possible is strongly advised.
* Prior history of organ transplant, including autologous stem cell transplant.
* Acute or sub-acute coronary syndromes within the last year, acute inflammatory heart disease, heart insufficiency NYHA > 2, or irreversible cardiac arrhythmias.
* A known impaired cardiac function defined as left ventricular ejection fraction (LVEF) < 50 % (or below the study site's lower limit of normal) as measured by MUGA or ECHO.
* Uncontrolled hypertensive disease; (systolic blood pressure (SBP) ≥160 or diastolic blood pressure (DBP) ≥100 mm Hg during two measurements).
* History or evidence of active autoimmune disease.
* Severe diabetic retinopathy (neoangiogenesis targeted by L19 outside the tumour).
* Major trauma, including oncologic surgery, but excluding smaller procedures like the placement of porth-à-cath or surgical biopsy, within 4 weeks prior to randomisation (neoangiogenesis targeted by L19 outside a tumour).
* Any underlying mental, medical or psychiatric condition which in the opinion of the investigator will make administration of study drug hazardous or hinder the interpretation of study results. Unstable or serious concurrent uncontrolled medical conditions.
* Pregnancy or breast feeding; it is well known that ED-B, the target of both L19IL2, is expressed in a variety of fetal tissues. Furthermore, anti-PD(L)1 treatment may increase the risk of immune-mediated disorders. Therefore, it will be contra-indicated for pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — trying to include 50% M/F in each group
Enrollment: 88 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 18 months after randomization of the last patient
  The main objective of the trial is to test the hypothesis that the combination of (SAB)R and L19-IL2 in patients with metastatic NSCLC will resulting in improved progression-free survival (PFS) compared to the SOC.

SECONDARY OUTCOMES:
Overall survival | 18 months after randomization of the last patient
  Assesment of the overall survival of the patient cohort.
Change in score of The EORTC quality of life questionnaire (QLQ) core module (C30) | baseline and at 3, 6, 9, 12, 15, 18, 21, 24 months after treatment
  The EORTC QLQ assesses health-related QoL of cancer patients; it consists of 30 items and covers 9 domains + 6 single symptoms. There are 5 functional scales: physical, role functioning, cognitive, emotional, social; 3 symptom scales: fatigue, pain, nausea + vomiting; a global health and QoL scale, and 6 single items. Each item has four response alternatives: 1) not at all, 2) a little 3) quite a bit 4) very much (score 1-4 with range 3); except for the global health-status/quality of life scale, which has options ranging from 1) very poor to 7) excellent (score 1-7, range 6). Answers are combined into dimensions and scores are linearly transformed into a score of 0 to 100 according to the scoring manual of the EORTC QoL group. For functional and global QoL scales, higher scores mean better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms. Scores are reported as mean and standard deviation. Scores will be used in multilevel-analysis.
Change in score of The EORTC quality of life questionnaire (QLQ) - Lung cancer module (LC13) | baseline and at 3, 6, 9, 12, 15, 18, 21, 24 months after treatment
  The EORTC QLQ-LC13 The Lung Cancer Module is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-LC13 incorporates one multi-item scale to assess dyspnoea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and haemoptysis. All items are scored 1 to 4, giving range = 3. After linear transformation scores range from 0 to100. A high score represents a high level of symptomatology or problems.
Change in score of The Euro Quality of Life - 5 dimensions - 5 levels (EQ-5D-5L) | baseline and at 3, 6, 9, 12, 15, 18, 21, 24 months after treatment
  EQ-5D-5L is a standardized instrument developed by the EuroQol Group as a measure of general health-related quality of life that can be used in a wide range of health conditions and treatments. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems (score 1-5). The scores for the five dimensions are combined into a 5-digit number that describes the patient's health state.
Change in score of The Euro Quality of Life (EQ) visual analogue scale (VAS) | baseline and at 3, 6, 9, 12, 15, 18, 21, 24 months after treatment
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale from 0-100. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Change in out of field radio-immune (OFRI) response | at 3, 6, 9, 12, 15, 18, 21, 24 months after treatment
  To assess the occurrence of an out of field radio-immune (OFRI) response, with a scan. Assessment will be based on the RECIST criteria.
Immunoresponse blood biomarkers by enzyme-linked immunosorbent assay (ELISA) | baseline and at 3, 6 and 9 months after treatment
  To perform correlative biomarker studies related to treatment response immunoresponse blood biomarkers will be measured: osteopontin (OPN), carbonic anhydrase IX (CA-IX)], interleukin-6 (IL-6), interleukin-8 (IL-8), C-reactive protein (CRP), carcinoembryonic antigen (CEA), cytokeratin fragment 21-1 (Cyfra 21-1), alpha-2-macroglobulin (α2M), serum interleukin-2 receptor (sIL2r), toll-like receptor 4 (TLR4), vascular endothelial growth factor (VEGF), extradomain-B fibronectin (EDB). This part of the study is exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastricht University
Locations (15):
- Belgium (4):
  - UCL St. Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - GZA Ziekenhuizen campus Sint-Augustinus, Wilrijk
- France (2):
  - Centre Oscar Lambret Lille, Lille
  - INSTITUT régional du CANCER MONTPELLIER - ICM - VAL d'AURELLE, Montpellier
- Germany (3):
  - University Hospital Carl Gustav Carus, Dresden
  - Klinikum der Universität Heidelberg, Heidelberg
  - University Hospital Tübingen, Tübingen
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS Università Cattolica del Sacro Cuore, Rome, Italy
- Netherlands (4):
  - Academisch Ziekenhuis Maastricht (Leading Centre), Maastricht, Limburg
  - AVL-NKI, Amsterdam
  - Radboud UMC Nijmegen, Nijmegen
  - Erasmus MC, Rotterdam
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Olivo Pimentel V, Marcus D, van der Wiel AM, Lieuwes NG, Biemans R, Lieverse RI, Neri D, Theys J, Yaromina A, Dubois LJ, Lambin P. Releasing the brakes of tumor immunity with anti-PD-L1 and pushing its accelerator with L19-IL2 cures poorly immunogenic tumors when combined with radiotherapy. J Immunother Cancer. 2021 Mar;9(3):e001764. doi: 10.1136/jitc-2020-001764. PMID 33688020
- [Derived] Lieverse RIY, Van Limbergen EJ, Oberije CJG, Troost EGC, Hadrup SR, Dingemans AC, Hendriks LEL, Eckert F, Hiley C, Dooms C, Lievens Y, de Jong MC, Bussink J, Geets X, Valentini V, Elia G, Neri D, Billiet C, Abdollahi A, Pasquier D, Boisselier P, Yaromina A, De Ruysscher D, Dubois LJ, Lambin P. Stereotactic ablative body radiotherapy (SABR) combined with immunotherapy (L19-IL2) versus standard of care in stage IV NSCLC patients, ImmunoSABR: a multicentre, randomised controlled open-label phase II trial. BMC Cancer. 2020 Jun 15;20(1):557. doi: 10.1186/s12885-020-07055-1. PMID 32539805
- See also: Website of ImmunoSABR trial — https://www.immunosabr.info/